CLINICAL TRIAL: NCT03526692
Title: Comparison of Effects Between SMR/Delta Ratio and beta1/Theta Ratio Neurofeedback Trainings for Older Adults With Mild Cognitive Impairment: A Protocol for a Randomized Controlled Trial
Brief Title: Neurofeedback Training for Older Adults With Mild Cognitive Impairment: a Protocol Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fabienne Marlats (Other)
Responsible Party: Sponsor-Investigator, Fabienne Marlats, PhD Candidate, Broca Hospital
Organization: Broca Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LUS1EEGNF
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment; Neurofeedback; electroencephalography; attention; memory
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: Comparison between three groups : two experimental groups and a control group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sensorimotor/delta NF training group (Experimental): Three interventions will be administered:
  * An electroencephalography recording (EEG) for 30 minutes.We will use an electrocap of 19 scalp locations according to the International 10-20 EEG placement system.
  * The second intervention is the neuropsychological assessments and questionnaires. They will be done in one session for approximately 2 hours.
  * The third intervention is the neurofeedback training sensorimotor/delta ratio that will be recorded at channel Cz according to the International 10-20 system.
  Interventions: Behavioral: Neurofeedback
- Beta1/theta NF training group (Experimental): Three interventions will be administered:
  * An electroencephalography recording (EEG) for 30 minutes.We will use an electrocap of 19 scalp locations according to the International 10-20 EEG placement system.
  * The second intervention is the neuropsychological assessments and questionnaires. They will be done in one session for approximately 2 hours.
  * The third intervention is the neurofeedback training Beta1/theta ratio that will be recorded at channel Fz according to the International 10-20 system.
  Interventions: Behavioral: Neurofeedback
- Control group (No Intervention): Three interventions will be administered:
  * An electroencephalography recording for 30 minutes.We will use an electrocap of 19 scalp locations according to the International 10-20 EEG placement system.
  * The second intervention is the neuropsychological assessments and questionnaires. They will be done in one session for approximately 2 hours.
  * The psychopedagogical care : Each session will be organized using the same video material than for the NF training sessions.

INTERVENTIONS:
Behavioral: Neurofeedback — Neurofeedback experiment will consist of 30 sessions of neurofeedback training, twice or three times a week during maximum 4 months. The two experimental groups will undergo questionnaires, EEG recording and neuropsychological assessments in three-time points, pre-training (T0), post-training (T1) and 3 months follow-up (T2). Electroencephalography will be recorded by a technician in EEGFor each participant, EEG power spectrum will be calculated in pre (T0) and post neurofeedback training/psycho-pedagogical care at T2 and T3.
  Other Names: Electroencephalography
  Arms: Beta1/theta NF training group; Sensorimotor/delta NF training group

SUMMARY:
This is a non-pharmacological study evaluating the effects of SMR/delta ratio and beta1/theta ratio neurofeedback trainings on cognitive performance and electrical brain activity in elderly with mild cognitive impairment.

DETAILED DESCRIPTION:
Older adults with Mild Cognitive Impairment (MCI) are at high risk to progress to Alzheimer's disease (AD). Slowing down effect of dementia by enhancing brain plasticity represents one of the most prominent challenges. Neurofeedback is one of the promising techniques that showed therapeutic efficacy and cognitive improvement in attention-deficit hyperactivity disorder, epilepsy, stroke. We aim to study the effects of two neurofeedback training protocols, SMR/delta ratio and beta1/theta ratio, on cognitive performances in older adults with Mild Cognitive Impairment and to assess whether MCI patients change in brain electrical activity in a resting state after training.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Mild Cognitive Impairment
* MMSE score >24
* Subjective memory complaint confirmed by an informant.
* Perform at/or below 1.5 standard deviations from the mean for age and education-matched norms on more than one of the neuropsychological tests.
* Preserve activity of daily living
* Absence of dementia.

Exclusion Criteria:

* Psychiatric and neurological disorders
* History of alcohol or other substance consumption

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Change on attention test, TMTB-TMA | Baseline Assessment in 2 weeks period before intervention, change from baseline at immediately after the end of the intervention and after 3-months follow-up
  assessment of the Trail Making Test B and A, calculation of subtraction

SECONDARY OUTCOMES:
Change on Rey Auditory Verbal Learning Test | Baseline assessment in 2 weeks period before intervention, change from baseline at immediately after the end of the intervention, and after 3-months follow-up
  Assessment of verbal learning in episodic memory

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie AR Rigaud, Professor, Principal Investigator — Broca University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marlats F, Bao G, Chevallier S, Boubaya M, Djabelkhir-Jemmi L, Wu YH, Lenoir H, Rigaud AS, Azabou E. SMR/Theta Neurofeedback Training Improves Cognitive Performance and EEG Activity in Elderly With Mild Cognitive Impairment: A Pilot Study. Front Aging Neurosci. 2020 Jun 16;12:147. doi: 10.3389/fnagi.2020.00147. eCollection 2020. PMID 32612522
- [Derived] Marlats F, Djabelkhir-Jemmi L, Azabou E, Boubaya M, Pouwels S, Rigaud AS. Comparison of effects between SMR/delta-ratio and beta1/theta-ratio neurofeedback training for older adults with Mild Cognitive Impairment: a protocol for a randomized controlled trial. Trials. 2019 Jan 29;20(1):88. doi: 10.1186/s13063-018-3170-x. PMID 30696475